CLINICAL TRIAL: NCT00999245
Title: Improving Pain Management and Outcomes With Various Strategies of Patient-Controlled Analgesia (PCA)
Brief Title: THE IMPROVE TRIAL: Improving Pain Management and Outcomes With Various Strategies of Patient-Controlled Analgesia (PCA)
Acronym: IMPROVE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Inability to meet target enrollment prior to ending of network in March 2011.
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 683; U10HL083721 (NIH)
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Demand / Low Infusion (Other): PCA dosing plan
  Interventions: Other: High Demand / Low Infusion
- Low Demand / High Infusion (Other): PCA plan for Low Demand / High Infusion
  Interventions: Other: PCA Dosing Plan

INTERVENTIONS:
Other: High Demand / Low Infusion — HDLI dosing plan will administer either morphine or hydromorphone using PCA. Dosing will be based on body weight.
  Other Names: HDLI
  Arms: High Demand / Low Infusion
Other: PCA Dosing Plan — LDHI dosing plan will administer either morphine ot hydromorphone using PCA. Dosing will be based on body weight.
  Other Names: LDHI
  Arms: Low Demand / High Infusion

SUMMARY:
Patient-Controlled Analgesia (PCA) means that the patient is in control of his/her pain medicine. In this study two (2) different treatment plans of Patient-Controlled Analgesia will be used to treat people with sickle cell disease who are admitted to the hospital for a pain crisis. The purpose of this study is to find out if one plan is better than the other in controlling sickle cell pain.

If you are eligible for the study, you will be assigned by chance (like flipping a coin) to either get a higher continuous amount of the pain medicine with a smaller amount for pain as you need it, OR to get a smaller continuous amount of pain medicine with a larger amount of pain medicine as you need it. You or your study doctor can not choose which plan you receive, and you will not be told which one you have been assigned to. The doctors and nurses taking care of you will know which plan you are assigned to so they can safely and effectively take care of your pain. Some members of the study team will not know which plan you are on.

We will give you morphine sulfate or hydromorphone (dilaudid) for your pain. These medicines are approved by the Food and Drug Administration (FDA) and have been used for a long time to relieve pain. If you have been treated for pain before with hydromorphone (dilaudid) and you prefer it to morphine, then you may choose to get it during the study. If you have not received hydromorphone (dilaudid) before or you do not have a preference then you will be given morphine for pain.

The pain medicine will be given through the IV in your arm. You will receive morphine or hydromorphone continuously through the IV and will also be able to use the PCA machine to give yourself extra pain medicine as you need it for pain. You will need to push a button to give yourself extra medicine for pain. The amount of pain medicine you get on these plans is based on how much you weigh.

DETAILED DESCRIPTION:
The following things will be done for the study:

1. Each day you are in the hospital someone from the study team who does not know your treatment assignment will come in 3 times during the day to ask you questions about your pain and how you are feeling. The doctors and nurses taking care of you will also do this as part of the routine care for your pain crisis. You will have your vital signs (blood pressure, heart rate, temperature) and oxygen level checked regularly as part of your routine care. The doctors and nurses may need to give you other medicines or do procedures that are not part of the study to take care of your pain crisis. They will talk with you about this. The doctors and nurses taking care of you while you are in the hospital will take care of you and treat your pain crisis just as they would do if you were not in this study. Being in this study will not interfere with the usual care and treatment you would receive.
2. Each day you are in the hospital a member of the study team will have you answer questions about your pain, any side effects you are having, and how well you are able to move around.
3. While you are in the hospital, you will wear an Actigraph Micro-Mini-Motion logger, a wristwatch type device that will keep track of how much you move around and how well you are sleeping. This will help us determine how well the treatment plan is relieving your pain level. You will wear the actigraph through Day 5 (Day 3 for children) of your hospital stay, or until you leave the hospital if you go home sooner.
4. Each day you are in the hospital you will have blood drawn to check how well your kidneys and liver are working. These blood tests will be done at the same time as your regular blood tests whenever possible. We will collect about 2 teaspoons of blood from you for the study each day you are in the hospital.
5. We will call you 3 days and 14 days after you leave the hospital. During these phone calls we will ask you questions about how you are feeling, the medications you are taking including those for pain, and any problems you have had since your discharge.

ELIGIBILITY:
Inclusion Criteria:

* Sickle Cell Disease: Hemoglobin diagnosis of SS (two copies of the hemoglobin S gene), SC (one copy of the hemoglobin S gene and one copy of the hemoglobin C gene), SD (one copy of the hemoglobin S gene and one copy of the hemoglobin D gene), or S-β thalassemia (β+ or β0)
* Male or female age ≥ 10 years.
* Typical vaso-occlusive pain that is not adequately controlled in an ambulatory or acute care setting and which is expected to require > 24 hours of hospital care.
* Pain Intensity Visual Analog (10 cm scale) score ≥ 4.5 cm, measured immediately after obtaining informed consent.
* Adults willing and able to give informed consent; parents willing and able to give permission for study participation by their children; minor subjects (ages 10-17) willing and able to provide assent.
* Ability to read/write English.

Exclusion Criteria:

* Medical Indication

  * Presence of significant liver disease (ALT > 3 times institutional upper limit of normal, or direct bilirubin > 0.8 mg/dl within preceding 3 months)
  * Presence of significant renal dysfunction (within preceding 3 months, creatinine ≥ 1.2 mg/dl for ages >18 yrs, or ages 10-18 yrs creatinine ≥ 1.0 mg/dl)
  * Oxygen saturation by pulse oximetry ≤ 92% on room air at study entry
  * Any other medical condition that renders the subject unable to or unlikely to complete the study or which would interfere with optimal participation in the study or which poses significant risk to the subject from study treatment including but not limited to:
  * Concurrent acute chest syndrome
  * Right upper quadrant pain
  * Symptomatic sleep apnea
  * Brain injury or doses of opioids that preclude potential subjects' capacity to give informed consent.
* Known (documented) hypersensitivity/intolerance to morphine and/or hydromorphone.
* Clinically significant opioid tolerance in the opinion of the investigator that precludes safe and/or effective dosing or requires, under current management, receiving the following long-acting oral opioids:

  * Methadone 40 mg/day
  * Sustained/Extended release oral morphine 120 mg /day
  * Oxycodone 80 mg/day
* Known pregnancy or currently breastfeeding.
* Poor venous access that in the investigator's judgment would preclude maintaining an IV throughout the admission.
* Currently participating in another research study.
* Previously randomized in the IMPROVE trial.
* Pain management in emergency department or Day Hospital ≥ 12 hours prior to decision to admit for inpatient care.
* Subject or physician preference for treatment with opioids other than morphine or hydromorphone.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To determine whether there is a difference in time to first occurrence of a large improvement in daily average pain intensity between a High Demand/Low Infusion (HDLI) dosing vs. Low Demand/High Infusion (LDHI) dosing for parenteral opioid. | Pain Intensity will be assessed 3 times a day between the hours of 7 AM and 7 PM on each day of the hospital stay

SECONDARY OUTCOMES:
The reduction in opioid usage as assessed by total (or parenteral) opioid usage during hospitalization for vaso-occlusive pain, as well as opioid usage by day of hospitalization. | up to Inpatient Day 3 for pediatric subjects and Inpatient Day 5 for adults or discharge whichever occurs first.
To compare the High Demand/Low Infusion (HDLI) vs. Low Demand/High Infusion (LDHI) treatment groups with respect to adverse events | Length of hospital stay
Assessment of opioid withdrawal symptoms as reported post discharge in two follow-up telephone calls | Follow up phone calls on Day 3 and Day 14 after discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Carlton Dampier, MD, Study Chair — Sickle Cell Disease Clinical Research Network; Wally Smith, MD, Study Chair — Sickle Cell Disease Clinical Research Network
Locations (28):
- United States (28):
  - Children's Hospital and Research Center, Oakland, California
  - Yale-New Haven Medical Center,, New Haven, Connecticut
  - A.I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Howard University Hospital, Washington D.C., District of Columbia
  - Emory University School of Medicine, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - University of Illinois Sickle Cell Center, Chicago, Illinois
  - Kosair Children's Hospital, Louisville, Kentucky
  - Children's Hospital at Sinai, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Interfaith Medical Center, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Ohio State University, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Virginia Commonwealth University Health Systems, Richmond, Virginia

REFERENCES:
- [Derived] Dampier CD, Smith WR, Wager CG, Kim HY, Bell MC, Miller ST, Weiner DL, Minniti CP, Krishnamurti L, Ataga KI, Eckman JR, Hsu LL, McClish D, McKinlay SM, Molokie R, Osunkwo I, Smith-Whitley K, Telen MJ; Sickle Cell Disease Clinical Research Network (SCDCRN). IMPROVE trial: a randomized controlled trial of patient-controlled analgesia for sickle cell painful episodes: rationale, design challenges, initial experience, and recommendations for future studies. Clin Trials. 2013 Apr;10(2):319-31. doi: 10.1177/1740774513475850. PMID 23539110